CLINICAL TRIAL: NCT05882409
Title: Effects of Education Given to University Students on Their Attitudes Towards Violence Against Women and Their Conflict and Awareness Levels
Brief Title: Education Given on Their Attitudes Towards Violence Against Women and Their Conflict
Acronym: violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Assoc. Prof. Dr., Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TR SIVAS 03
Record Dates: First submitted 2023-05-10; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: University Students; Attitudes; Conflict; Education; Women; Violence; Awareness
Keywords: Awareness; Conflic; Education; Student; Violence against women
MeSH Terms: conditions — Behavior | interventions — Educational Status; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): In the experimental groups the education whose content (definition and importance of violence and conflict, violence against women, the cycle of violence, who is at risk for violence, characteristics of perpetrators and the victims of violence, types of violence against women, consequences of violence and conflict on individuals, legal aspects of violence, positive coping with violence and conflict, empowering women against violence, conflict resolution) was prepared by the researcher in line with the adult education principles and pertinent literature was given in the school prepared for education beforehand. In accordance with the adult education principles, the students were educated in groups of 12-15 people. During the education, methods such as narration, discussion, question-answer, brainstorming, problem solving and summarizing, data shows, brochures, posters and visual materials were used. The duration of the education lasted 30-40 minutes.
  Interventions: Behavioral: Education
- Standard of care Group (No Intervention): The control group did not receive any treatment.

INTERVENTIONS:
Behavioral: Education — Education covers women's education on violence, conflict and awareness.
  Other Names: Control Group
  Arms: Education group

SUMMARY:
Introduction: Violence against women is the violation of human rights faced by women of all ages, cultures and education levels everywhere. It can be experienced in many different ways, either individually or socially.

Aim: The study was conducted to investigate the effects of education given to university students on their attitudes towards violence against women, and their conflict and awareness levels.

DETAILED DESCRIPTION:
Methods: The sample of this randomized controlled experimental study comprised 87 (experimental group=45; control group=42) university students studying in health-related fields. The students in the experimental group received in one session education on violence against women and conflict, whereas the students in the control group did not receive any education. The study data were collected with the Personal Information Form, Attitudes towards Violence Scale among University Students, and Conflict and Violent Awareness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Women who lived in the city center,
* University students
* Studying in health-related fields
* Women who volunteered to participate in the study

Exclusion Criteria:

* Being a man
* Training other than health-related fields
* Those who do not live in the city center
* Involuntary

Ages: 18 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Attitudes towards Violence Scale among University Students | 5 months
  The scale consisted of 52 items, scored between 1-5 and the total score is calculated
Conflict and Violent Awareness Scale | 5 months
  The scale consisted of 27 items, scored between 1-5 and the total score is calculated

CONTACTS AND LOCATIONS:
Overall Officials: Sukran E Ertekin Pinar, Principal Investigator — Cumhuriyet University
Locations (1):
- Sukran Ertekin Pinar, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No